CLINICAL TRIAL: NCT00282035
Title: An RCT to Determine if APBI, Utilizing 3D CRT, is as Effective as Whole Breast Irradiation Following Breast Conserving Surgery in Women With Ductal Carcinoma in Situ or Invasive Breast Cancer With Negative Axillary Lymph Nodes
Brief Title: RAPID: Randomized Trial of Accelerated Partial Breast Irradiation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Canadian Breast Cancer Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OCOG-2005-RAPID; CIHR Grant Number: MCT-78567 (Other Grant/Funding Number: CIHR)
Record Dates: First submitted 2006-01-23; First posted 2006-01-25 (Estimated); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Breast Cancer
Keywords: breast cancer; breast tumour; DCIS; female; breast conserving surgery; irradiation; whole breast irradiation; 3D CRT accelerated partial breast irradiation; cosmetic outcome; quality of life
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- APBI utilizing 3D-CRT radiation (Experimental): Accelerated partial breast irradiation utilizing 3D-CRT
  Interventions: Radiation: APBI utilizing 3D-CRT radiation
- Whole breast irradiation (Other): Whole breast irradiation
  Interventions: Radiation: Whole breast irradiation

INTERVENTIONS:
Radiation: APBI utilizing 3D-CRT radiation — Accelerated partial breast irradiation utilizing 3D-CRT
  Arms: APBI utilizing 3D-CRT radiation
Radiation: Whole breast irradiation — Whole breast irradiation
  Arms: Whole breast irradiation

SUMMARY:
To determine if Accelerated Partial Breast Irradiation, using 3D CRT, is as effective as Whole Breast Irradiation following breast conserving surgery in women with an new histological diagnosis of ductal carcinoma in situ only or invasive breast cancer without evidence of metastatic disease. Effectiveness will be determined by the rate of ipsilateral breast tumour recurrence.

General objective is to improve the convenience and quality of life of female patients who receive breast irradiation.

DETAILED DESCRIPTION:
Following breast conserving surgery or on completion of chemotherapy, patients will be stratified according to age, tumour histology, tumour size, adjuvant hormonal therapy and clinical centre. Patients will be allocated to receive either whole breast irradiation or 3D CRT accelerated partial breast irradiation.

Radiation therapy will be administered as soon as possible following the healing of the surgical incision (3-4 weeks) and within 12 weeks if the patient is not treated with chemotherapy. If the patient is treated with chemotherapy, radiation therapy will begin after 2 weeks and not beyond 8 weeks after the last dose of chemotherapy.

Patients treated with whole breast irradiation will receive a total dose of 42.5 Gy in 16 fractions, given on a daily basis, over a time period of 22 days. Patients with large breast size are permitted to receive a total dose of 50 Gy in 25 fractions, given on a daily basis, over a time period of 35 days. Boost irradiation is permitted in patients treated with whole breast irradiation. Boost irradiation of 10 Gy/4-5 fractions daily over a time period of 4-7 days is permitted for patients deemed at moderate to high risk of local recurrence as per local cancer centre guidelines.

Patients treated with 3D CRT accelerated partial breast irradiation will receive a total dose of 38.5 Gy in 10 fractions, delivered twice a day, over a time period of 5-8 days. Each daily dose must be separated by 6-8 hours.

Patients will be followed indefinitely and assessed formally at 6 and 12 months after the date of randomization and then on a yearly basis. Patients will be assessed for acute and late radiation toxicity, cardiac toxicity, recurrent disease, new primary cancer, cosmetic outcome, quality of life and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* 1a. Female patient with a new histological diagnosis of DCIS only. OR

  1b. Female patient with a new histological diagnosis of invasive carcinoma of the breast and no evidence of metastatic disease.

  2. Treated by BCS with microscopically clear resection margins for invasive and non-invasive disease (or no residual disease on re- excision).

  3. Negative axillary node involvement including micrometastasis <= 0.2mm or positive cells only identified by IHC as determined either by: (i) sentinel node biopsy (ii) axillary node dissection or (iii) clinical exam for patients with DCIS only

Exclusion Criteria:

* 1. Age < 40 years.

  2. A known deleterious mutation in BRCA 1 and/or BRCA 2.

  3. Tumour size > 3 cm in greatest diameter on pathological examination (including both the invasive and non-invasive component).

  4. Tumour histology limited to lobular carcinoma only.

  5. History of cancer:
  * Patients with another active malignancy or malignancy treated < 5 years prior to randomization are excluded.
  * Patients with a prior diagnosis of invasive or non-invasive breast cancer in either breast are excluded regardless of disease free interval. Patients with concurrent invasive or non-invasive contralateral breast cancer are also excluded.
  * Patients with prior or concurrent basal cell or squamous cell skin cancers are eligible for the trial.

    6. More than one primary tumour in different quadrants of the same breast.

    7. Previous irradiation to the ipsilateral breast that would preclude whole breast irradiation.

    8. Presence of an ipsilateral breast implant or pacemaker.

    9. Serious non-malignant disease (e.g. cardiovascular, pulmonary, systemic lupus erythematosus (SLE), scleroderma) which would preclude definitive radiation treatment.

    10. Estrogen receptor status (ER) not known.

    11. For patients not treated with adjuvant chemotherapy: unable to commence radiation therapy within 12 weeks of the last surgical procedure on the breast.

    12. For patients treated with adjuvant chemotherapy: unable to commence within 8 weeks of the last dose of chemotherapy.

    13. Currently pregnant or lactating.

    14. Psychiatric or addictive disorders which would preclude obtaining informed consent or adherence to protocol.

    15. Geographic inaccessibility for follow-up.

    16. Inability to localize surgical cavity on CT (i.e., no evidence of surgical clips or seroma).

    17. Inability to adequately plan the patient for the experimental technique.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2135 (Actual)
Dates: Start 2006-01; Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
ipsilateral breast tumour recurrence defined as recurrent invasive or in situ cancer in the ipsilateral breast including the axillary tail. | ongoing throughout study
  ipsilateral breast tumour recurrence

SECONDARY OUTCOMES:
adverse cosmetic outcome | evaluated at 1, 3, 5, 7 and 10 years
  adverse cosmetic outcome
disease free survival | ongoing throughout study
  disease free survival
event free survival | ongoing throughout study
  event free survival
overall survival | ongoing throughout study
  overall survival
radiation toxicity | ongoing throughout study
  radiation toxicity
quality of life based on questionnaire responses | ongoing throughout study
  quality of life
cost effectiveness | end of study
  cost effectiveness

CONTACTS AND LOCATIONS:
Overall Officials: Tim Whelan, MD, Principal Investigator — Ontario Clinical Oncology Group / Juravinski Cancer Centre; Ivo Olivotto, MD, Principal Investigator — British Columbia Cancer Agency - Vancouver Island Centre; Mark Levine, MD, Study Director — Ontario Clinical Oncology Group (OCOG)
Locations (33):
- Australia (4):
  - Peter MacCallum Cancer Centre, Bendigo, Victoria
  - Peter MacCallum Cancer Centre, Box Hill, Victoria
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
  - Peter MacCallum Cancer Centre - Monash Medical Centre Moorabbin, Melbourne, Victoria
- Canada (28):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BC Cancer Agency - Abbotsford Centre, Abbotsford, British Columbia
  - British Columbia Cancer Agency - Centre for the Southern Interior, Kelowna, British Columbia
  - British Columbia Cancer Agency - Fraser Valley Centre, Surrey, British Columbia
  - British Columbia Cancer Agency - Vancouver Centre, Vancouver, British Columbia
  - British Columbia Cancer Agency - Vancouver Island Centre, Vancouver, British Columbia
  - Cancer Care Manitoba, Winnipeg, Manitoba
  - Atlantic Health Sciences Corporation, Saint John, New Brunswick
  - QE II HSC - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Brantford General Hospital, Brantford, Ontario
  - Northeastern Regional Cancer Centre, Greater Sudbury, Ontario
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Grand River Regional Cancer Centre, Kitchener, Ontario
  - London Regional Cancer Centre, London, Ontario
  - Credit Valley Hospital - Carlo Fidani Peel Regional Cancer Center, Mississauga, Ontario
  - Durham Regional Cancer Centre - Lakeridge Health Corporation, Oshawa, Ontario
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Irving Greenberg Family Cancer Centre, Ottawa, Ontario
  - Niagara Health System, St. Catharines, Ontario
  - Princess Margaret Hospital - University Health Network, Toronto, Ontario
  - Windsor Regional Cancer centre, Windsor, Ontario
  - CHUS - Hopital Fleurimont, Fleurimont, Quebec
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - CHUM - Hospital Notre Dame, Montreal, Quebec
  - McGill University - Montreal General Hospital, Montreal, Quebec
  - McGill University - Jewish General Hospital, Montreal, Quebec
  - CHUQ, L'Hotel Dieu de Quebec, Québec, Quebec
- Auckland City Hospital, Auckland, Auckland, New Zealand

REFERENCES:
- [Derived] Whelan TJ, Julian JA, Berrang TS, Kim DH, Germain I, Nichol AM, Akra M, Lavertu S, Germain F, Fyles A, Trotter T, Perera FE, Balkwill S, Chafe S, McGowan T, Muanza T, Beckham WA, Chua BH, Gu CS, Levine MN, Olivotto IA; RAPID Trial Investigators. External beam accelerated partial breast irradiation versus whole breast irradiation after breast conserving surgery in women with ductal carcinoma in situ and node-negative breast cancer (RAPID): a randomised controlled trial. Lancet. 2019 Dec 14;394(10215):2165-2172. doi: 10.1016/S0140-6736(19)32515-2. Epub 2019 Dec 5. PMID 31813635